CLINICAL TRIAL: NCT02530307
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled 21-Day Treatment Study, Including an fMRI Sub-Study, to Evaluate the Effect of HT-3951 on Upper Extremity Motor Function Following Ischemic Stroke
Brief Title: HT-3951 vs. Placebo in Stroke Rehabilitation
Acronym: RESTORE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative
Sponsor: Dart NeuroScience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-3951-201
Record Dates: First submitted 2015-08-06; First posted 2015-08-21 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Ischemic Stroke
Keywords: Stroke,; Rehabilitation; Ischemic; fMRI
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HT-3951 (15mg) (Experimental): HT-3951 capsules administered once daily
  Interventions: Drug: HT-3951
- Placebo (Placebo Comparator): Placebo capsules administered once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HT-3951
  Arms: HT-3951 (15mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel group outpatient study that will utilize standard stroke rehabilitation outcome measures, as well as fMRI techniques in a subset of subjects, to evaluate the effect of HT-3951 on motor recovery and behavior in medically stable subjects following ischemic stroke.

ELIGIBILITY:
Main Inclusion Criteria:

* Age range between 21 to 85 years, inclusive, at the Screening Visit
* Subjects who have experienced an ischemic stroke documented by CT or MRI resulting in an upper extremity deficit that, in the opinion of the Investigator, warrants the need for rehabilitation therapy
* Medically stable subjects who are able to be randomized to study medication beginning between ≥ 2 and ≤ 52 weeks post-stroke
* Subjects who have initiated, are undergoing, have completed or agree to begin physical or occupational rehabilitation for at least 2 weeks prior to study Day 1.
* Mild to moderate unilateral upper extremity motor impairment characterized by FMA-EU score of > 18
* Modified Rankin Scale score of 1 to 4

Main Exclusion Criteria:

* History of stroke within 6 months prior to the subject's current episode of ischemic stroke (History of transient ischemic attacks or ischemic stroke (nonhemorrhagic) more than 6 months prior to the current ischemic stroke are acceptable.)
* Subjects with unresolved upper or lower motor deficits (e.g., range of motion or strength deficits) from any prior stroke
* Significant hemorrhagic stroke
* Any history of seizure disorder or a spontaneous seizure that had occurred at any time after the stroke
* Apraxia that, in the Investigator's opinion, would likely reduce the ability of the subject to participate in the study or confound study outcome measures
* Moderate to severe aphasia and/or severe language deficits
* Severe sensory loss in affected hand
* Moderate to severe hemispatial neglect or anosognosia involving the affected arm
* Absent proprioception at the elbow or shoulder joints
* Excessive spasticity in the affected elbow, defined as a score of greater than or equal to 3 on the Modified Ashworth Spasticity scale (MAS)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity, Part A-D | 21-days
Index Finger-Tapping Frequency Test | 21-days
Nine-Hole Peg Test | 21-days
Hand Grip Strength Dynamometer Test | 21-days
Arm Motor Ability Test-9 | 21-days
Stroke Impact Scale (hand domain) | 21-days
Somatosensory evoked potential (if available) | 21-days

SECONDARY OUTCOMES:
Two-Minute Walk Test | 21-days
Behavioral, neural activity and motor network connectivity levels, using functional MRI | 21-days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Perera, MD, Study Director — Dart NeuroScience, LLC
Locations (18):
- United States (18):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Downey, California
  - Glendale, California
  - Loma Linda, California
  - Orlando, Florida
  - Chicago, Illinois
  - Grand Rapids, Michigan
  - Kansas City, Missouri
  - West Orange, New Jersey
  - New York, New York
  - White Plains, New York
  - Charlotte, North Carolina
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Elkins Park, Pennsylvania
  - Dallas, Texas
  - Houston, Texas